CLINICAL TRIAL: NCT05386862
Title: Wayne Warrior CAnnabis Research and Education: Naturalistic Observation and Harm Reduction
Brief Title: Warrior CARE: Naturalistic Observation and Harm Reduction
Acronym: NOC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study protocol was revised, which required closing it and submitting a new application. Since recruitment launched for this protocol, no participants were enrolled and run in this study protocol.
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Leslie Lundahl, Associate Professor, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Warrior CARE: NOC
Record Dates: First submitted 2022-04-28; First posted 2022-05-23 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Post Traumatic Stress Disorder; Cannabis Use; Suicide
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naturalistic Group (No Intervention): This group will followed as they follow their naturalistic cannabis use.
- THC Reduction Group (Experimental): This group will be asked to reduce the THC content and increase CBD content of their cannabis products to study the effect of PTSD symptom severity.
  Interventions: Behavioral: Reduce THC Use

INTERVENTIONS:
Behavioral: Reduce THC Use — Reducing THC concentrations and increasing CBD to reduce PTSD symptom severity
  Arms: THC Reduction Group

SUMMARY:
This study is looking at therapeutic potential of reducing Tetrahydrocannabinol (THC) levels in regular cannabis smokers using contingency management (CM) intervention in a U.S. veteran population with post-traumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
In this trial, the investigators will recruit veterans with post-traumatic stress disorder (PTSD) who report using cannabis. Veterans will be assigned (via participant self-selection) into either a naturalistic group that will be followed as the participants continue to use cannabis as they normally do (observation only), or into a "THC (tetrahydrocannabinol) reduction group" in which veterans are asked to switch from their typical cannabis product to using a lower THC/higher Cannabidiol (CBD) product; adherence to this switch will be incentivized using a behavioral intervention called contingency management (CM).

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent, IQ Score >80,
* served in branch of the US armed forces, report using cannabis,
* report using cannabis (at least 4x/month)
* test positive for THC in urine drug screen,
* meet DSM-5 criteria for PTSD w/ Sx of at least 6 months duration

Exclusion Criteria:

* urine drug screen positive for any other drugs
* any clinically significant medical problems,
* any current or past serious psychotic or bipolar disorder diagnosis as determined by SCID-5
* at immediate high risk for suicide based on the C-SSRS
* current SUD other than Nicotine Use Disorder, Alcohol (mild or moderate) and Cannabis Use Disorder
* seeking treatment for Cannabis Use Disorder

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Change in Clinician-Administered PTSD Scale for DSM-5 Total Severity Score (CAPS-5) | Baseline, 3, 6, 12 months post baseline
  Assessing change in PTSD symptom severity from baseline, to 3, 6, and 12 months post baseline. A decrease in the CAPS-5 assessment indicates less PTSD symptoms endorsed and a better outcome. Minimum score is 0, maximum score is 20 for PTSD subtotals.
Change in Post-Traumatic Stress Disorder Symptom Checklist for DSM-5 (PCL-5) | Baseline, every 2 weeks for 12 weeks, 3, 6, 12 months post baseline
  Assessing change in PTSD symptom and severity over time. This scale is completed by the participants and a lower score indicates less PTSD symptoms and better study outcomes. Maximum score is 80 and minimum score is 20.
Change in Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline, 3, 6, 12 months post baseline
  Suicide ideation, intensity, and behavior assessment. This is a clinical interview to assess suicide severity. Reduction in suicide related behaviors represents a better study outcome.
Change in Suicide Behavior Questionnaire - Revised (SBQ-R) | Baseline, every 2 weeks for 12 weeks, 3, 6, 12 months post baseline
  Suicide ideation, intensity, and behavior assessment completed by participants. Scores range from 3 to 18, with lower score representing better study outcome.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory-II | Baseline, every 2 weeks for 12 weeks, 3, 6, 12 months post baseline
  Self report depression checklist. Beck Depression Inventory-II scores range from 0 to 63 and lower score represent better outcome.
Change in State Trait Anxiety Inventory Form Y | Baseline, every 2 weeks for 12 weeks, 3, 6, 12 months post baseline
  Anxiety symptom checklists ranging from from 20 to 80. Lower scores on this measures represents better study outcome.
Change in California Verbal Learning Test | Baseline, 3, 6, 12 months post baseline
  Verbal memory task that will be used to measure the change in executive function over time.
Change in Wisconsin Card Sort Task | Baseline, 3, 6, 12 months post baseline
  Computer task that will be used to measure the change in executive function over time.
Change in Iowa Gambling Task | Baseline, 3, 6, 12 months post baseline
  Computer task that measure the change in decision making over time.
Change in General Health Survey (Short form 36) | Baseline, 3, 6, 12 months post baseline
  General health questionnaire to assess change in general health outcomes over time. General health survey is scored from 0 to 100 with a higher score denoting better study outcomes.
Change in Quality of Life Inventory | Baseline, 3, 6, 12 months post baseline
  Quality of Life assessment to examine change in quality of life over time. Quality of life inventory is scored from 16 to 112, higher score indicating better study outcome.
Change in Brief Pain Inventory | Baseline, 3, 6, 12 months post baseline
  Brief pain inventory asks participants identify areas on their body causing pain and rate the severity. Less pain symptoms over time represent a better study outcome.
Exploratory analysis of genetic markers associated with endocannabinoid system | Baseline
  DNA analysis to examine genetic markers associated with the endocannabinoid system. The genetic data will be collected from blood samples during baseline. Data will be grouped based on genetic variants of proteins within the endocannabinoid system to identify genetic differences in response to the treatment trial.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Lundahl, PhD, Principal Investigator — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olenick M, Flowers M, Diaz VJ. US veterans and their unique issues: enhancing health care professional awareness. Adv Med Educ Pract. 2015 Dec 1;6:635-9. doi: 10.2147/AMEP.S89479. eCollection 2015. PMID 26664252
- [Background] Boden MT, Babson KA, Vujanovic AA, Short NA, Bonn-Miller MO. Posttraumatic stress disorder and cannabis use characteristics among military veterans with cannabis dependence. Am J Addict. 2013 May-Jun;22(3):277-84. doi: 10.1111/j.1521-0391.2012.12018.x. PMID 23617872
- [Background] Adkisson K, Cunningham KC, Dedert EA, Dennis MF, Calhoun PS, Elbogen EB, Beckham JC, Kimbrel NA. Cannabis Use Disorder and Post-Deployment Suicide Attempts in Iraq/Afghanistan-Era Veterans. Arch Suicide Res. 2019 Oct-Dec;23(4):678-687. doi: 10.1080/13811118.2018.1488638. Epub 2018 Nov 17. PMID 29952737
- [Background] Hill MN, Bierer LM, Makotkine I, Golier JA, Galea S, McEwen BS, Hillard CJ, Yehuda R. Reductions in circulating endocannabinoid levels in individuals with post-traumatic stress disorder following exposure to the World Trade Center attacks. Psychoneuroendocrinology. 2013 Dec;38(12):2952-61. doi: 10.1016/j.psyneuen.2013.08.004. Epub 2013 Sep 10. PMID 24035186
- [Background] Hill MN, Miller GE, Ho WS, Gorzalka BB, Hillard CJ. Serum endocannabinoid content is altered in females with depressive disorders: a preliminary report. Pharmacopsychiatry. 2008 Mar;41(2):48-53. doi: 10.1055/s-2007-993211. PMID 18311684
- [Background] deRoon-Cassini TA, Stollenwerk TM, Beatka M, Hillard CJ. Meet Your Stress Management Professionals: The Endocannabinoids. Trends Mol Med. 2020 Oct;26(10):953-968. doi: 10.1016/j.molmed.2020.07.002. Epub 2020 Aug 28. PMID 32868170
- [Background] Abizaid A, Merali Z, Anisman H. Cannabis: A potential efficacious intervention for PTSD or simply snake oil? J Psychiatry Neurosci. 2019 Mar 1;44(2):75-78. doi: 10.1503/jpn.190021. No abstract available. PMID 30810022
- [Background] Zachary RA (1991) Shipley Institute of Living Scale: revised manual. Los Angeles: Western Psychological Services
- [Background] First MB, Williams JBW, Karg RS, Spitzer RL (2015) User's Guide for the Structured Clinical Interview for DSM-5 Disorders, Research Version (SCID-5-RV). Arlington, VA, American Psychiatric Association
- [Background] Weathers, F.W., et al., The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). 2013, Washington DC: National Center for PTSD.
- [Background] Weathers, F.W., Litz, B.T., Keane, T.M., Palmieri, P.A., Marx, B.P., & Schnurr, P.P. (2013). The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov.
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Osman A, Bagge CL, Gutierrez PM, Konick LC, Kopper BA, Barrios FX. The Suicidal Behaviors Questionnaire-Revised (SBQ-R): validation with clinical and nonclinical samples. Assessment. 2001 Dec;8(4):443-54. doi: 10.1177/107319110100800409. PMID 11785588
- [Background] Beck, A.T., Steer, R.A., & Brown, G.K. (1996). Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation.
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Wechsler, D. (2009). Wechsler Memory Scale - 4th Edition. Pearson Assessments.
- [Background] BERG EA. A simple objective technique for measuring flexibility in thinking. J Gen Psychol. 1948 Jul;39:15-22. doi: 10.1080/00221309.1948.9918159. No abstract available. PMID 18889466
- [Background] Milner, B. (1963). Effects of different brain lesions on card sorting. Archives of Neurology, 9, 90-100.
- [Background] Bechara A, Damasio H, Tranel D, Damasio AR. Deciding advantageously before knowing the advantageous strategy. Science. 1997 Feb 28;275(5304):1293-5. doi: 10.1126/science.275.5304.1293. PMID 9036851
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Frisch, M.B., Cornell, J., Villanueva, M. & Retzlaff, P.J. (1992). Clinical validation of the quality of life inventory: A measure of life satisfaction for treatment planning and outcome assessment. Psychological Assessment, 4, 92-101.
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Marczylo TH, Lam PM, Nallendran V, Taylor AH, Konje JC. A solid-phase method for the extraction and measurement of anandamide from multiple human biomatrices. Anal Biochem. 2009 Jan 1;384(1):106-13. doi: 10.1016/j.ab.2008.08.040. Epub 2008 Sep 18. PMID 18823934
- [Background] Matias I, Gatta-Cherifi B, Tabarin A, Clark S, Leste-Lasserre T, Marsicano G, Piazza PV, Cota D. Endocannabinoids measurement in human saliva as potential biomarker of obesity. PLoS One. 2012;7(7):e42399. doi: 10.1371/journal.pone.0042399. Epub 2012 Jul 31. PMID 22860123
- [Background] Maples-Keller JL, Rauch SAM, Jovanovic T, Yasinski CW, Goodnight JM, Sherrill A, Black K, Michopoulos V, Dunlop BW, Rothbaum BO, Norrholm SD. Changes in trauma-potentiated startle, skin conductance, and heart rate within prolonged exposure therapy for PTSD in high and low treatment responders. J Anxiety Disord. 2019 Dec;68:102147. doi: 10.1016/j.janxdis.2019.102147. Epub 2019 Sep 21. PMID 31669786
- [Background] Norr AM, Smolenski DJ, Reger GM. Effects of prolonged exposure and virtual reality exposure on suicidal ideation in active duty soldiers: An examination of potential mechanisms. J Psychiatr Res. 2018 Aug;103:69-74. doi: 10.1016/j.jpsychires.2018.05.009. Epub 2018 May 12. PMID 29783077
- [Background] Haney M, Ward AS, Comer SD, Foltin RW, Fischman MW. Abstinence symptoms following smoked marijuana in humans. Psychopharmacology (Berl). 1999 Feb;141(4):395-404. doi: 10.1007/s002130050849. PMID 10090647
- [Background] Haney M, Hart CL, Ward AS, Foltin RW. Nefazodone decreases anxiety during marijuana withdrawal in humans. Psychopharmacology (Berl). 2003 Jan;165(2):157-65. doi: 10.1007/s00213-002-1210-3. Epub 2002 Nov 19. PMID 12439626
- [Background] Petry NM, Alessi SM, Ledgerwood DM. Contingency management delivered by community therapists in outpatient settings. Drug Alcohol Depend. 2012 Apr 1;122(1-2):86-92. doi: 10.1016/j.drugalcdep.2011.09.015. Epub 2011 Oct 5. PMID 21981991
- [Background] Petry NM, Alessi SM, Ledgerwood DM. A randomized trial of contingency management delivered by community therapists. J Consult Clin Psychol. 2012 Apr;80(2):286-98. doi: 10.1037/a0026826. Epub 2012 Jan 16. PMID 22250852
- [Background] Ellis JD, Struble CA, Fodor MC, Cairncross M, Lundahl LH, Ledgerwood DM. Contingency management for individuals with chronic health conditions: A systematic review and meta-analysis of randomized controlled trials. Behav Res Ther. 2021 Jan;136:103781. doi: 10.1016/j.brat.2020.103781. Epub 2020 Nov 30. PMID 33302054
- [Background] Ledgerwood DM, Arfken CL, Petry NM, Alessi SM. Prize contingency management for smoking cessation: a randomized trial. Drug Alcohol Depend. 2014 Jul 1;140:208-12. doi: 10.1016/j.drugalcdep.2014.03.032. Epub 2014 Apr 13. PMID 24793364
- [Background] Reid HH, Ledgerwood DM. Depressive symptoms affect changes in nicotine withdrawal and smoking urges throughout smoking cessation treatment: Preliminary results. Addict Res Theory. 2016;24(1):48-53. doi: 10.3109/16066359.2015.1060967. Epub 2015 Jun 26. PMID 27547173
- [Background] Bilgin M, Bindila L, Graessler J, Shevchenko A. Quantitative profiling of endocannabinoids in lipoproteins by LC-MS/MS. Anal Bioanal Chem. 2015 Jul;407(17):5125-31. doi: 10.1007/s00216-015-8559-8. Epub 2015 Mar 18. PMID 25782872
- [Background] Gachet MS, Rhyn P, Bosch OG, Quednow BB, Gertsch J. A quantitiative LC-MS/MS method for the measurement of arachidonic acid, prostanoids, endocannabinoids, N-acylethanolamines and steroids in human plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2015 Jan 22;976-977:6-18. doi: 10.1016/j.jchromb.2014.11.001. Epub 2014 Nov 18. PMID 25436483
- [Background] Marczylo TH, Lam PM, Amoako AA, Konje JC. Anandamide levels in human female reproductive tissues: solid-phase extraction and measurement by ultraperformance liquid chromatography tandem mass spectrometry. Anal Biochem. 2010 May 15;400(2):155-62. doi: 10.1016/j.ab.2009.12.025. Epub 2009 Dec 22. PMID 20026294
- [Background] Watkins BA, Kim J, Kenny A, Pedersen TL, Pappan KL, Newman JW. Circulating levels of endocannabinoids and oxylipins altered by dietary lipids in older women are likely associated with previously identified gene targets. Biochim Biophys Acta. 2016 Nov;1861(11):1693-1704. doi: 10.1016/j.bbalip.2016.07.007. Epub 2016 Jul 22. PMID 27452639
- [Background] McDougle DR, Watson JE, Abdeen AA, Adili R, Caputo MP, Krapf JE, Johnson RW, Kilian KA, Holinstat M, Das A. Anti-inflammatory omega-3 endocannabinoid epoxides. Proc Natl Acad Sci U S A. 2017 Jul 25;114(30):E6034-E6043. doi: 10.1073/pnas.1610325114. Epub 2017 Jul 7. PMID 28687674
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865